CLINICAL TRIAL: NCT06335043
Title: Personalized Pharmacotherapy Using Pharmacogenetics in Veterans Seeking Treatment for Mental Health
Brief Title: Personalized Pharmacotherapy Using Pharmacogenetics in Veterans
Acronym: PGx
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Don Richardson, Scientific Director, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 119245
Record Dates: First submitted 2024-03-13; First posted 2024-03-28 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Pharmacogenetic Testing to Determine Pharmacological Treatment in PTSD

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Mental Health Provider (No Intervention): Mental health provider's thoughts on pharmacogenetic testing for treatment planning and changes to treatment planning.
- Patient with Pharmacogenetic Testing (Experimental): For patient participants who opt-in to pharmacogenetic testing, a report summarizing the pharmacogenetic testing results will be sent to each patient participants' respective mental health provider.
  Interventions: Genetic: Pharmacogenetics Testing
- Patient without Pharmacogenetic Testing (No Intervention): For patient participants who opt-out to pharmacogenetic testing will be followed to see if treatment course is maintained.

INTERVENTIONS:
Genetic: Pharmacogenetics Testing — Genetic test to determine individual genetic compatibility with multiple pharmaceutical drug classes to determine best outcomes for prescription drug treatment.
  Arms: Patient with Pharmacogenetic Testing

SUMMARY:
This study is an observational clinical trial aimed at to evaluate the use of pharmacogenetic testing (PGx) for mental health treatment in members and Veterans of the CAF and RCMP patient population as well as the attitudes of both St. Joseph's OSI Clinic Psychiatrists and patients towards PGx. Both OSI Clinic Psychiatrists participants and patient participants will be administered a brief demographic survey in addition to a survey examining their views on, and current knowledge of PGx. Patient participants will have an opportunity to opt-in to or opt-out of receiving PGx. For patient participants who opt-in to PGx (PGx-guided treatment group), a report summarizing the PGx results will be sent to each patient participants' respective OSI Clinic Psychiatrist, alongside a questionnaire that captures the OSI Clinic Psychiatrist participant's treatment planning and changes to treatment planning. Where applicable, past treatment data from patient participants acquired at the St. Joseph's OSI Clinic will be used to identify the number of prior medication changes. Patient participants who opt-out of PGx but continue to receive pharmacologic care at the St. Joseph's OSI Clinic will act as a standard care comparator treatment group. Patient participant's outcomes including PTSD, depression and anxiety severity, and medication-related side effects, will be assessed until the patient participant is discharged from the OSI Clinic or after 24 weeks, whichever comes first. All patient participants, regardless of their study treatment group, will have their symptomatology collected via standard care data collection protocol (Client Reported Outcomes Monitoring Information System (CROMIS) and electronic medical records (EMR)); a self-report assessing the presence of side effects will be completed via Lawson REDCap. OSI Clinic Psychiatrist participants and patient participants will be asked to complete a virtual exit interview at the end of their participation.

ELIGIBILITY:
Inclusion Criteria:

* Provider participant:

  * Are at least 18 years of age;
  * Speak and write English;
  * Currently working as an OSI Clinic Psychiatrist at the London St. Joseph's OSI Clinic.

    * Psychiatrist with an active caseload of patients being treated for OSIs.
* Patient participant:

  * Veteran (patient) CAF or RCMP member;
  * Are at least 18 years of age;
  * Are a current patient at the London St. Joseph's OSI Clinic;
  * Current diagnosis of an OSI;
  * Speak and write English;
  * Consents to the use of CROMIS data for the purpose of this study; and
  * Consents to the use of prior OSI Clinic data for research purposes (if you have been a patient at the OSI Clinic prior to this study, the research team will use past OSI Clinic data to observe changes over time).

Exclusion Criteria:

* Participants (provider or patients) who are unable to, or do not, provide informed consent for participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 155 (Estimated)
Dates: Start 2024-04-25 (Actual); Primary Completion 2027-04-25 (Estimated); Study Completion 2027-04-25 (Estimated)

PRIMARY OUTCOMES:
PHQ-9 - Patient Health Questionnaire 9 | 5 minutes
  Objectifies degree of depression severity
GAD-7 - General Anxiety Disorder-7 | 5 minutes
  Measures severity of anxiety
PCL-5 - Posttraumatic Stress Disorder Checklist - 5 | 5 minutes
  A 20-item self-report tool that corresponds to the 20 symptoms listed in the DSM-V
OQ-45 - Outcome Questionnaire 45 | 10 minutes
  A 45-item multiple-choice self-report inventory used to measure psychotherapy progress in adult patients
Pharmacological Side Effect Measure | 10 minutes
  To determine if the participant is experiencing any new or worsening or continuing side effects related to prescription medications
Electronic Medical Record Extraction Measure | 10 minutes
  To determine trial and error attempts with pharmacological prescriptions in an attempt to minimize and/or control symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- MacDonald Franklin OSI Research and Innovation Centre, London, Ontario, Canada